CLINICAL TRIAL: NCT00872482
Title: A Randomized, Phase II, Double-Blind Study of Nimotuzumab Plus Whole-Brain Radiation Therapy (WBRT) Compared With WBRT Alone in Patients With Brain Metastases From Non-Small Cell Lung Cancer
Brief Title: A Study of Nimotuzumab in Combination With Radiation Therapy in Patients With Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to low enrollment
Sponsor: YM BioSciences (Industry)
Collaborators: CIMYM BioSciences (Other)
Responsible Party: Wendy Chapman, Vice President, Clinical Operations, YM BioSciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YMB1000-018
Record Dates: First submitted 2009-03-26; First posted 2009-03-31 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; NSCLC; Brain metastases; nimotuzumab; TheraCIM; h-R3; Radiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nimotuzumab (200 mg fixed dose) will be administered by the intravenous route weekly during WBRT and following WBRT. Radiotherapy will consist of 30 Gy, in 10 fractions of 3 Gy/day.
  Interventions: Drug: nimotuzumab
- 2 (Placebo Comparator): A placebo will be administered by the intravenous route weekly during WBRT and following WBRT.
  Radiotherapy will consist of 30 Gy, in 10 fractions of 3 Gy/day.
  Interventions: Drug: nimotuzumab

INTERVENTIONS:
Drug: nimotuzumab — Nimotuzumab (200 mg fixed dose) will be administered by the intravenous route weekly during WBRT and following WBRT Radiotherapy will consist of 30 Gy, in 10 fractions of 3 Gy/day.

SUMMARY:
This is a randomized, Phase II study designed to investigate Nimotuzumab plus whole-brain radiation therapy (WBRT)and to compare it rith WBRT alone in patients with brain metastases from non-small cell lung cancer (NSCLC). The purpose of the study is to assess the efficacy of nimotuzumab in combination with WBRT.

DETAILED DESCRIPTION:
A phase II, randomized, controlled, double blinded and multicenter study with 2 arms, administering the study drug during radiotherapy and following radiotherapy until disease progression, unacceptable toxicity or at the discretion of the physician. Randomization will be done 2:1 (experimental:control). Chemotherapy can be added before documented disease progression at the discretion of the physician.

The primary objective is to assess the efficacy of Nimotuzumab in combination with WBRT. The primary endpoint is intracranial disease progression over 6 months.

The secondary endpoints are overall survival (OS); time to neurologic progression (TNP) or death with evidence of neurologic progression; OS rate at 6 months; time to intracranial disease progression; and time to overall progression.

Tissue samples and serum will be collected for future correlative studies.

All the images will be centrally reviewed at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Providing a written informed consent (see Appendix A);
* Age ≥18 years;
* Histologic or cytologic confirmed diagnosis of NSCLC of any epithelial type (squamous, adenocarcinoma, large cell, or other);
* At least one newly diagnosed measurable metastatic lesion from NSCLC in the brain;
* Patient had initial diagnosis of brain metastases by image, within 8 weeks of registration
* KPS ≥70;
* Absolute neutrophil count ≥ 1500/mm³;
* Platelet count ≥ 50,000/mm³;
* Serum creatinine ≤2.0 mg/dL;
* Serum transaminases ≤2 x the upper limit of normal (ULN);
* Total serum bilirubin ≤2 x ULN;
* And a lactate dehydrogenase (LDH) level ≤1.3 x ULN.

Exclusion Criteria:

* Pregnancy, lactation or parturition within the previous 30 days (fertile female or male patients should practice contraception);
* Prior WBRT, brain metastases resection with no other measurable lesion remaining;
* Extracranial metastases in two or more organs;
* Known leptomeningeal or subarachnoid tumor spread;
* Plan to use radiosurgery or radiation boost after completion of WBRT;
* Plan to use chemotherapy or any other systemic antineoplastic modality during WBRT;
* Previous use of an anti-EGFR drug;
* Participation in another ongoing therapeutic trial;
* Presence of known HIV seropositivity, severe comorbidities, or other malignant neoplasm within 5 years (except adequately treated basal- or squamous-cell carcinoma of skin or in situ carcinoma of the uterine cervix);
* Hypersensitivity or allergy to any of the drugs to be administered in this study;
* Inability or unwillingness to complete the required assessments;
* Geographic inaccessibility for treatment or follow-up evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Phase II: efficacy.Withhold of intracranial progression at 2, 4 and 6 months in comparison with control arm. Patients will be assessed by lab tests, MRI,neurologic examination | weekly infusions during radiotherapy and following radiotherapy until disease progression, unacceptable toxicity or withdrawal of consent.

SECONDARY OUTCOMES:
Overall survival (OS); time to neurologic progression (TNP) or death with evidence of neurologic progression; OS rate at 6 months; time to intracranial disease progression; and time to overall progression. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Brade, M.D., Principal Investigator — Assitant Professor, Department of Radiation Oncology, University of Toronto
Locations (15):
- United States (3):
  - Florida Cancer Institute - New Hope, New Port Richey, Florida
  - Park Nicollet Institute - Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Overlake Hospital Medical Center, Bellevue, Washington
- Canada (8):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Royal Victoria Hospital, Barrie, Ontario
  - London Regional Cancer Center, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hotel Dieu Hospital, Québec, Quebec
- Hospital Clínico Quirúrgico Hermanos Ameijeiras, Centro Habana, La Habana, Cuba
- Pakistan (2):
  - Hameed Latif Hospital, Lahore (HLH), Town, Lahore
  - Nuclear Medicine and Radiation Oncology Institute (NORI), Islamabad
- Severance Hospital, Seoul, South Korea